CLINICAL TRIAL: NCT06807996
Title: Effects of Zinc Supplementation on Patients With Elevated Glycemic Status: A Randomized Double-blind Placebo-controlled Clinical Trial
Brief Title: Effects of Zinc Supplementation on Patients With Elevated Glycemic Status
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhilei Shan (Other)
Responsible Party: Sponsor-Investigator, Zhilei Shan, Professor, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: S235
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-03

CONDITIONS: Elevated Blood Glucose
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Zinc supplementation (Experimental): zinc-enriched yeast capsule, 15mg/d
  Interventions: Dietary Supplement: Zinc-enriched yeast capsule
- Edible yeast placebo (Placebo Comparator): Edible yeast placebo capsule, 15mg/d
  Interventions: Dietary Supplement: Edible yeast placebo capsule

INTERVENTIONS:
Dietary Supplement: Zinc-enriched yeast capsule — Daily zinc supplementation: zinc-enriched yeast capsules (15 mg) for a total of 6 months.
  Arms: Zinc supplementation
Dietary Supplement: Edible yeast placebo capsule — Daily edible yeast placebo capsules (not zinc-enriched) (15 mg) for a total of 6 months.
  Arms: Edible yeast placebo

SUMMARY:
The goal of this randomized, double-blind, placebo-controlled study included patients with elevated glycemic status is to investigate whether zinc supplementation (4mg per day) has beneficial effects on controlling blood glucose.

DETAILED DESCRIPTION:
The goal of this randomized, double-blind, placebo-controlled study included patients with elevated glycemic status is to investigate whether zinc supplementation (4mg per day) has beneficial effects on controlling blood glucose.

About 124 patients aged 18 years or older, had resided locally for at least one year, with elevated glycemic status will be enrolled in the study. Patients with elevated glycemic status are defined as meeting any of the following criteria:

1. Fasting blood glucose ≥ 6.1 mmol/L;
2. Glycated hemoglobin (HbA1c) ≥ 5.7%;
3. Oral glucose tolerance test (OGTT) 2-hour or postprandial blood glucose ≥ 7.8 mmol/L;
4. Patients with previously diagnosed type 2 diabetes with stable drug hypoglycemic treatment and blood glucose controlled well.

Eligible participants will be assigned by chance to one of two groups: (1) daily zinc supplementation: zinc-enriched yeast capsules (4 mg); (2) daily edible yeast placebo capsules (not zinc-enriched) (4mg). Randomization will be conducted.

At enrollment, baseline questionnaires are designed to collect data on sociodemographic factors, lifestyle habits, health status, and medical conditions. Participants in both groups will take one capsule that contained either Zinc-enriched yeast or edible yeast placebo each day until the end of the intervention period.

Participants will be followed up two times (3 months and 6 months post-intervention), and receive a single stage-specific dosage at any given follow-up time. During each follow-up visit, participants will complete a questionnaire survey, a 3-day 24-hour dietary recall, and undergo physical measurements. Blood, urine, and stool samples will also be obtained in the study center, fasting blood glucose, HbA1c and other biochemical indicators will also be detected at the same time.

The primary outcomes, including fasting blood glucose and HbA1c will be measured using blood samples. Secondary outcomes in this study include changes in blood lipids (such as total cholesterol, triglycerides, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol), trends in plasma zinc levels, inflammatory factors, oxidative stress indexes, other blood indicators and liver and kidney function indicators. Data will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Fasting blood glucose ≥ 6.1 mmol /L;
2. HBA1c ≥ 5.7%;
3. OGTT 2-hour or postprandial blood glucose ≥ 7.8 mmol/L;
4. Patients with previously diagnosed type 2 diabetes with stable drug hypoglycemic treatment and blood glucose controlled well.

Exclusion Criteria:

1. Age < 18 years, or currently pregnant;
2. Individuals with severe obesity, thyroid disease, cardiovascular or cerebrovascular diseases, or other serious health conditions;
3. Individuals with a previous diagnosis of type 2 diabetes currently receiving insulin therapy;
4. Individuals who have taken zinc-related supplements within three months prior to baseline inclusion;
5. Individuals using other nutritional supplements or with poor lifestyle habits;
6. Individuals with unstable body weight in the past three months (fluctuations > 5 kg);
7. Individuals with a history of major surgery within the past three months or planned major surgery within the next month;
8. Individuals allergic to the intervention materials;
9. Individuals who did not adhere to the prescribed consumption of the study product, affecting efficacy or safety assessment;
10. Individuals with positive urinary protein or serum creatinine greater than 1.2 times the upper limit of normal (men: serum creatinine > 133.2 μmol/L, women: serum creatinine > 97.2 μmol/L) at screening;
11. Individuals with elevated alanine aminotransferase (ALT) levels at screening (men: ALT > 50 U/L, women: ALT > 35 U/L).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Concentration of fasting blood glucose (FBG) | 0 week, 12th week, and 24th week in the intervention period
  Concentration of FBG, measured in mmol/L
Glycated hemoglobin (HbA1c) | 0 week, 12th week, and 24th week in the intervention period
  Concentration of HbA1c, measured in the percentage of hemoglobin

SECONDARY OUTCOMES:
Concentration of fasting plasma insulin (FPI) | 0 week, 12th week, and 24th week in the intervention period
  Concentration of FPI, measured in μIU/mL
Concentration of plasma c-peptide | 0 week, 12th week, and 24th week in the intervention period
  Concentration of plasma c-peptide, measured in nmol/L
Homeostatic model assessment of insulin resistance (HOMA-IR) | 0 week, 12th week, and 24th week in the intervention period
  HOMA-IR can be calculated as (FPI [μU/mL] × FBG [mmol/L]) / 22.5
Homeostatic model assessment of β-cell function (HOMA-β) | 0 week, 12th week, and 24th week in the intervention period
  HOMA-β is calculated as (20 × FPI [μU/mL]) / (FBG [mmol/L] - 0.195)
Homeostatic model assessment of insulin sensitivity (HOMA-S) | 0 week, 12th week, and 24th week in the intervention period
  HOMA-S is calculated as 1 / HOMA-IR
Concentration of blood lipids | 0 week, 12th week, and 24th week in the intervention period
  Concentration of blood lipids: total cholesterol, triglycerides, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol, measured in mmol/L
Concentration of C-reactive protein (CRP) | 0 week, 12th week, and 24th week in the intervention period
  Concentration of CRP, measured in mg/dL
Concentration of interleukin-6 (IL-6) | 0 week, 12th week, and 24th week in the intervention period
  Concentration of IL-6, measured in pg/mL
Concentration of malondialdehyde (MDA) | 0 week, 12th week, and 24th week in the intervention period
  Concentration of MDA, measured in μmol/L
Activity of Cu-Zn superoxide dismutase (SOD) | 0 week, 12th week, and 24th week in the intervention period
  Activity of Cu-Zn SOD, measured in U/mL
Concentration of homocysteine (HCY) | 0 week, 12th week, and 24th week in the intervention period
  Homocysteine (HCY) [μmol/L]
Concentration of plasma albumin (ALB) | 0 week, 12th week, and 24th week in the intervention period
  Concentration of ALB, measured in g/dL
Concentration of plasma creatinine | 0 week, 12th week, and 24th week in the intervention period
  Concentration of plasma creatinine, measured in μmol/L
Concentration of plasma zinc | 0 week, 12th week, and 24th week in the intervention period
  Concentration of plasma zinc concentrations, measured in mg/dL

IPD SHARING:
Plan to Share IPD: No